| A Group-Based Walking Study to Enhance Physical Activity Among Older Adults: The Role of Social Engagement |
|---|

Informed Consent Form
NCT03803085

Document Date: 7/22/2019

## **WeChat Study Informed Consent**

This research study, which is conducted by the Boston Roybal Center for Active Lifestyle Interventions at Brandeis University, is about using the app, WeChat to help you increase your physical activity by walking.

This study will take place over the course of 4 weeks. The study can be one at home; you do not need to come to the university. At the beginning and end we will ask you to fill out a series of questionnaires. Completing the questionnaires at each of the two occasions (at the beginning and end of the study) should take about 30 minutes each time, and you can do this in your own home at times that are convenient for you. You will download WeChat on your smart phone, which you may keep upon completion of the study. You will be sent reminders on your smartphone each day. At the end of the 4-week period and then 1 month after, you will be asked again to fill out the questionnaires, at a convenient time.

WeChat is a cross-platform communication service that combines the popular features of Facebook and WhatsApp. We will evaluate the WeRun function in WeChat to further foster peer support while increasing motivation, exercise self-efficacy, social contact with other older adults, and well-being. Any risks involved in this study are minimal and no greater than those encountered in everyday life. It is possible, although unlikely, that some participants may experience an injury or become physically fatigued from engaging in an increased amount of activity.

The direct personal benefits associated with participating in this study include using the WeChat to keep upon completion of the study. You will also receive one \$25 giftcard at the beginning and another \$25 giftcard at the completion of the study.

If you increase your physical activity you may also experience benefits to your overall health. The information collected by the researchers will be entirely confidential and will be used for research purposes only. Your name will not be used in any reports and all of your responses, including the information provided by internet, phone calls, and the app will be identified by a number and not your name. Data for all participants will be combined and analyzed as a group. Therefore, we will not be able to give you specific feedback about your individual results. Upon request, we will be happy to send you a summary of the overall research findings when they are available.

Your participation in this study is voluntary; and you are completely free to withdraw from the study at any time or to refuse to answer any questions, or to decline participation in any component of the study. If you do not complete the study, you will still be able to keep the app.

By signing below, you state that you have heard and understand the explanation of this study and freely consent to participate in it; that you understand that your participation is voluntary; and that you are completely free to withdraw from the study at any time or to refuse to answer any questions, or to decline participation in any component in the study.

By signing below, you agree that all questions you may have had about the study have been explained to your full satisfaction. If you have further questions about the study, you may contact the Principal Investigator, Margie Lachman, or her research assistant at the Lifespan Lab 781 736 3284. If you have questions about your rights as a research subject please contact the Brandeis Institutional Review Board at irb@brandeis.edu or 781-736-8133.

| Participant's name (please print): | |
|------------------------------------|-------|
| Participant's signature: | Date: |
| Researcher's signature: | Date: |

Please sign and return this form using the enclosed stamped and addressed envelope to:
Boston Roybal Center for Active Lifestyle Interventions Lifespan Lab
Brandeis University
Brown Social Sciences Building Psychology Department MS 062
415 South Street
Waltham, MA 02454